CLINICAL TRIAL: NCT01406080
Title: Single-blinded, Multicenter, Randomized, Comparative Study of Efficacy and Safety of Adapalene Gel 0.3% Versus Tretinoin Emollient Cream 0.05% in the Treatment of Cutaneous Photoaging.
Brief Title: A Comparative Study of Adapalene Gel,0.3% Versus Tretinoin Emollient Cream, 0.05% for the Treatment of Photoaging
Acronym: FOTEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma Brasil Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BR.10.002
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2016-01

CONDITIONS: Photoaging; Photodamage
Keywords: Photoaging; Photodamage; Adapalene; Differin
MeSH Terms: interventions — Adapalene; Tretinoin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adapalene (Active Comparator): Differin® gel 0.3% (adapalene Gel 0,3%)
  Interventions: Drug: Adapalene
- Tretinoin (Active Comparator): Tretinoin 0,05% emollient cream
  Interventions: Drug: Tretinoin

INTERVENTIONS:
Drug: Adapalene — Apply approximately 1 gram of Differin 0.3% every night on the entire face, except near the eye region.
  Other Names: Differin® Gel 0.3%; Adapalene Gel 0.3%
  Arms: Adapalene
Drug: Tretinoin — Apply approximately 1 gram of Tretinoin emollient cream 0.05% every night on the entire face, except near the eye region.
  Other Names: Tretinoin emollient cream 0,05%
  Arms: Tretinoin

SUMMARY:
The purpose of this study is to:

1. Evaluate the efficacy of Adapalene gel 0.3% compared to Tretinoin Emollient cream 0.05%, reducing signs of cutaneous photoageing, measured trough photonumeric scale evaluation, investigator evaluation of global response to treatment and subject's evaluation of improvement.
2. Evaluate the safety and tolerability of Adapalene Gel 0.3%, compared to Tretinoin Emollient cream 0.05% during 24 weeks of treatment.

The study has the clinical hypothesis that Adapalene Gel 0.3% is as effective as Tretinoin Emollient cream 0.05% in the treatment of cutaneous photoaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at least some score on periorbital or frontal wrinkle or melanosis and at maximum a "Severe" score on any of the criteria considered in evaluating cutaneous photoaging extension, based on the table for assessing Cutaneous Photoaging Extent;
* Male and female patients aged at least 35 years and maximum of 55 years, with skin phototype of I to IV, according to the T.B. Fitzpatrick's scale;
* Individuals who have mild to moderate cutaneous photoaging, i.e., score 2-6 in the overall assessment of cutaneous photoaging, based on the Griffiths scale;
* If female, individuals who cannot get pregnant (defined as post-menopausal the lack of menstrual bleeding for one year - or have undergone bilateral tubal ligation, hysterectomy or bilateral oophorectomy) or, if in childbearing age, patients who underwent urine pregnancy test with negative results. Patients should be using an appropriate contraceptive method. In the case of oral contraceptives, the use must have been started at least one month before the study or 12 months in case of pills containing cyproterone. Patients should maintain the same contraceptive during the study and 1 additional month after completion;
* For subjects under treatment for a concomitant medical condition, type and dose must be stable for at least three months prior to study entry (at least one year, in the case of hormone replacement therapy) and should not change during the study. These drugs do not include the excluded drugs cited in exclusion criterion;
* Individuals able to avoid prolonged sun exposure, especially on the face during the study period and willing to use the proper techniques to avoid the sun, including the use of sunscreen provided during the study;
* Individuals able to follow the study instructions and who are willing to complete all required visits;
* Individuals who have signed the informed consent form before any study procedures;

Exclusion Criteria:

* Patients who have participated in another clinical trial for less than 30 days;
* Pregnant women, nursing mothers or women attempting to conceive;
* Female patients who started hormone replacement therapy for less than one year before entering the study;
* Individuals with a condition or who are in a situation that, in the opinion of the investigator, may put the objective of the study at risk, confound the results or even interfere with the individual participation. These include, but are not limited to:

  1. Individuals with other facial skin disorders or dermatosis (scars, inflammatory acne, etc.) that can interfere with the clinical evaluation;
  2. Patients with a history of treatment for photoaging using ablative laser technologies (such as carbon dioxide and Erbium: YAG) and / or non-ablative (Nd: YAG, Fractionated Erbium Glass, Diode, Infrared Light, Intense Pulsed Light, Radiofrequency, Pulsed Dye Laser), dermabrasion, medium or deep chemical peeling on face;
  3. Individuals diagnosed with skin cancer (squamous cell carcinoma, melanoma) in the last 3 months prior to study entry;
  4. Individuals not willing to refrain from any cosmetic procedure during the study period (e.g. other types of chemical peelings, microdermabrasion, etc.);
  5. Individuals with significant medical history, concomitant disease or condition in which the investigator believes that participation in the study is not propitious;
* Patients with known sensitivity to retinoids or to any component of the study products;
* Patients with a diagnosis or history of keloids;
* Patients without the minimum wash-out period for the following treatments:

  1. 2 weeks for topical alpha- hydroxy acid, glycolic acid, salicylic acid, lactic acid, betahydroxy acid on the face.
  2. 2 weeks for topical products containing vitamin A, ascorbic acid, vitamin E on the face.
  3. 2 weeks for topical corticosteroids.
  4. 4 weeks for systemic corticosteroids.
  5. 3 months for topical retinoids.
  6. 1 year for oral retinoids.
* Patients who underwent superficial chemical peelings, microdermabrasion or exfoliation on the face in the last 3 months;
* Patients who applied botulinum toxin or soft tissue fillers for facial rejuvenation in the last 6 months and do not agree on not using these products during the study;
* Patients self-identified as "sensitive skin";
* Patients who are not willing or able to attend the study visits;

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Assessing the extent of Cutaneous Photoaging at the end of treatment. | Baseline to week 24
  Evaluation of Cutaneous Photoaging Extension at the end of treatment: the signs of cutaneous photoaging are evaluated by means of reduction of at least one point in any one of the following parameters: periorbital wrinkles, ephelides / melanosis, forehead wrinkles, tactile roughness (texture) and actinic keratosis.

SECONDARY OUTCOMES:
Global Assessment of photoaging, based on the Griffiths photonumeric scale. | week 24
  The evaluator, blinded to the treatment, will assess the global degree of photoaging of the patient in all visits, based on photographic images of the Griffiths scale consisted of 5 categories (Periorbital Wrinkles, Ephelides / melanosis, Forehead Wrinkles, Tactile roughness (texture), Actinic Keratosis. These were evaluated on a scale from 0 - 4 (0 = Absent, 1 = Minimal, 2 = Mild, 3 = Moderate and 4 = Severe) with 0 being best and 4 being worst.
Assessing the extent of Cutaneous Photoaging at each visit. | week 24
  The absolute values and changes of the Evaluation of Cutaneous Photoaging Extent in relation to baseline will be summarized by using frequency tables and at each visit and the groups will be compared.
Evaluation of Improvement by the Investigator at Week 12 | week 12
  The evaluator, blinded to the treatment, will evaluate the improvement of the photoaging signs at week 12 using the scale 5 = important response, 4 = near complete response (≈ 90% improvement), 3 = marked response (≈ 75% improvement), 2 = moderate response (≈ 50% improvement), 1 = mild response (≈ 25% improvement), 0 = No answer, -1= Worsening.
Evaluation of Improvement by the Investigator at Week 24 | Week 24
  The evaluator, blinded to the treatment, will evaluate the improvement of the photoaging signs at week 12 using the scale 5 = important response, 4 = near complete response (≈ 90% improvement), 3 = marked response (≈ 75% improvement), 2 = moderate response (≈ 50% improvement), 1 = mild response (≈ 25% improvement), 0 = No answer, -1= Worsening.
Subject Assessment of improvement at week 24. | week 24
  Patients will evaluate the improvement perceived at week 24 using the following scale:0 = Improves hard to notice, 1 = A very small improvement, 2 = Small improvement, 3 = Moderate improvement, 4 = Major improvements.
Anatomical-pathological assessment | week 24
  The difference between the treatment arms in epidermal thickness and 7.7 in the thickness of the granular layer will be detect at week 24.
Digital morphometric assessment. | week 24
  The thickness of the stratum corneum, granular layer and the epithelium will be estimated

CONTACTS AND LOCATIONS:
Overall Officials: Ananda Quadros Campos, Study Director — Galderma Brasil Lltda; Edileia Bagatin, Principal Investigator — Universidade Federal de São Paulo
Locations (4):
- Brazil (4):
  - Centro de Dermatologia Dona Libania, Fortaleza, Ceará
  - Santa Casa de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital de Clínicas da Universidade Federal do Paraná, Curitiba, Paraná
  - Universidade Federal de São Paulo - UNIFESP - UNICCO, São Paulo, São Paulo